CLINICAL TRIAL: NCT04389047
Title: Comparison of Two Mechanical Ventilation Strategies on Tissue Oxygenization of Patients Undergoing Bariatric Surgery
Brief Title: Comparison of Two Mechanical Ventilation Modes on Oxygenisation
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01.02.2013-228
Record Dates: First submitted 2020-01-20; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Bariatric Surgery Candidate; Mechanical Ventilation; Hypoxia; Tissue Damage
Keywords: bariatric surgery, tissue oxygenization, ventilation
MeSH Terms: conditions — Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison the effect of two different mechanical ventilation modes on tissue oxygenization.

DETAILED DESCRIPTION:
Aim of the study is to evaluate and compare the effects of two different mechanical ventilation modes as Volume Controlled Mechanical Ventilation (VCV) and Pressure Controlled Mechanical Ventilation (PCV) on non invasive tissue oxygenization levels of patients who scheduled for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients with Body Mass Index 35 - 50 kg/m2 Patients classified as American Society of Anesthesiologist (ASA) 1-2-3 classification Patients elected for Bariatric surgery

Exclusion Criteria:

Patients who wants to reject of study participation Patients who has any surgical complication during the surgery period Patients with decompensated cardiac failure Patients with Moderate or Severe obstructive/restrictive lung disease Patients with Reynaud disease Patients with Buerger phenomena Patients whıo has Intraoperative airway pressure more than 45 cmH2O Patients who had previous thoracic surgery Patients with Negative Modified Allen test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population involves the elective bariatric surgery patients who have body mass index between 35 and 50 kg/m2.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2013-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Oxygenization | peroperative 0. minute - 15. minute - 30. minute - 45. minute - 60. minute
  Peroperative Non invazive technique of Superficial Tissue Oxygenization
Oxygenization-2 | post operative 1. hour - 4. hour - 8. hour - 12. hour - 24.hour
  Post operative Non invazive technique of Superficial Tissue Oxygenization
Arterial blood gas analysis | Peroperative 0. minute - 30. minute - 60. minute
  Lactate, Ph, Arterial oxygen pressure, Arterial Carbondioxide pressure, Oxygen Saturation
Arterial blood gas analysis-2 | post operative 1.hour - 4. hour - 8. hour - 12. hour - 24.hour
  Lactate, Ph, Arterial oxygen pressure, Arterial Carbondioxide pressure, Oxygen Saturation
Peripheral oxygen saturation | peroperative 0. minute - 15. minute - 30. minute - 45. minute - 60. minute
  Peripheral Oxygen Saturation (SpO2)
Peripheral oxygen saturation-2 | post operative 1.hour - 4. hour - 8. hour - 12. hour - 24.hour
  Peripheral Oxygen Saturation (SpO2)

SECONDARY OUTCOMES:
Peroperative hemodynamic measurements | peroperative 0. minute - 15. minute - 30. minute - 45. minute - 60. minute
  Heart rate, Mean Arterial Blood Pressure
Postoperative hemodynamic measurements | post operative 1.hour - 4. hour - 8. hour - 12. hour - 24.hour
  Heart rate, Mean Arterial Blood Pressure
Carbondioxide | peroperative 15. minute - 30. minute - 45. minute - 60. minute
  End tidal Carbondioxide measurement

IPD SHARING:
Plan to Share IPD: Undecided